CLINICAL TRIAL: NCT02775409
Title: Prospective Trial of Subcutaneous Versus Subpectoral 2-Staged Implant-Based Breast Reconstruction
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Minh-Doan Nguyen, Assistant Professor of Plastic Surgery, Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 16-000539
Record Dates: First submitted 2016-05-13; First posted 2016-05-17 (Estimated); Last update posted 2021-12-30 (Actual); Status verified 2021-12

CONDITIONS: Breast Reconstruction Following Mastectomy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Subcutaneous (Active Comparator): Subcutaneous placement of tissue expander
  Interventions: Procedure: Subcutaneous placement
- Submuscular (Active Comparator): Submuscular placement of tissue expander
  Interventions: Procedure: Submuscular placement

INTERVENTIONS:
Procedure: Subcutaneous placement — The tissue expander will be placed above the muscle.
  Arms: Subcutaneous
Procedure: Submuscular placement — The tissue expander will be placed below the muscle
  Arms: Submuscular

SUMMARY:
This study is for women scheduled to have immediate breast reconstruction following mastectomy using a tissue expander. The primary purpose of this study is to learn whether there are differences in the outcome between placing the tissue expander above the muscle or below the muscle. The study will evaluate pain, wellbeing, and overall satisfaction with reconstruction. A secondary purpose is to learn whether there are differences in complications and costs between the two locations.

ELIGIBILITY:
Inclusion Criteria:

1. Women at least 18 years of age, who will undergo immediate unilateral or bilateral implant-based breast reconstruction following therapeutic skin-sparing or nipple-sparing mastectomy.
2. Women at least 18 years of age, who will undergo immediate bilateral implant-based breast reconstruction following risk-reduction (prophylactic) skin-sparing or nipple-sparing mastectomy.

Exclusion Criteria:

1. Subjects who are unable to read or speak English.
2. Patients desiring autologous reconstruction.
3. BMI >40.
4. History of radiation therapy to the breast(s), e.g. history of breast conservation therapy.
5. Current nicotine and/or tobacco use.
6. Documented diagnosis of chronic pain.
7. Women who are pregnant or breast-feeding *
8. Women who decline the use of acellular dermal matrix (ADM).
9. Surgeon decision not to proceed with tissue expander reconstruction.
10. Women undergoing single stage (straight to implant) reconstruction.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2016-05-01 (Actual); Primary Completion 2020-02-06 (Actual); Study Completion 2020-02-06 (Actual)

PRIMARY OUTCOMES:
Change in patient satisfaction | Baseline, Year 3
  Difference in patient satisfaction between the two groups using the physical well being scale.

CONTACTS AND LOCATIONS:
Overall Officials: Minh-Doan Nguyen, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: Yes
Present/publish results at professional meetings/journals

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials